CLINICAL TRIAL: NCT07252713
Title: Complex Rehabilitation Technology Enabled Physical Activity for Children With Motor Delays Via Telehealth in Natural Environments
Acronym: CP-MOVES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Director, PEARL Lab, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20251878
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy (CP); Motor Disability; Motor Delay
Keywords: Assistive Device; Stander; Physical Activity; Sedentary; Parent; Physical Therapy; Rehabilitation; Digital Health; Telehealth; Wearable Sensors
MeSH Terms: conditions — Cerebral Palsy; Psychomotor Disorders; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth-delivered parent coaching intervention in adaptive stander use (Experimental): Children will receive an adaptive stander and complete 30-minute sessions 3 times per week for 8 weeks. One session per week will be telehealth-delivered with a study researcher.
  Interventions: Behavioral: Stander Use

INTERVENTIONS:
Behavioral: Stander Use — The intervention includes 8 weeks of adaptive standing training delivered via telehealth with PT parent-coaching (1 telehealth session/week + 2 parent-led practice sessions/week). Sessions are 30 minutes, 3x/ week. Participants are provided a stander, sized to their age and body size for use during the study.

SUMMARY:
The primary goal of CP-MOVES is to evaluate 1) the preliminary efficacy of a telehealth-delivered, parent coaching intervention in the use of adaptive standers, on physical activity, sleep, and endurance in young children with severe motor delays and 2) on physical activity, sedentary time, resting heart rate, and perceived stress in parents.

The main questions we aim to answer include:

1. Do measures of physiological fitness and sleep in children with severe motor delays (i.e., unable to stand without support) change after a therapist-directed, parent-delivered intervention using telehealth and adaptive standers?
2. Do parents report any changes in their child's endurance, participation, or quality of life OR parent stress following intervention?

Children ages 1-6 years old with severe motor delay and one parent will:

1. Complete three 30 minute sessions of standing in an adapted stander per week for 8 weeks. One session per week will be completed with a physical therapist, delivered through telehealth and two sessions per week will be completed as a home program with the parent and child (no therapist or telehealth).
2. Wear activity tracker sensors on the wrist(s) and waist for one-week before and after treatment.
3. Complete questionnaires about the child's endurance, participation, and quality of life and the parent's stress, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Child age 1-6 years with CP or other severe motor delay (GMFCS IV-V);
* Unable to stand without external support;
* Parent willing and able to participate;
* Internet access for telehealth;
* Live within 100 miles of lab or travel for device provision,
* One parent is fluent in English.

Exclusion Criteria:

* Inability to participate in telehealth
* Parent/caregiver unable to participate

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Wearable sensor physical activity data: Vector Magnitude | From enrollment to end of 8-week treatment period
  Vector Magnitude is a measure of moderate to vigorous physical activity measured in G-Force units. To be measured pre/post in parent and child.
Wearable sensor physical activity data: Daily Activity Counts | From enrollment to end of 8-week treatment period
  Wearable sensor outcomes measured in parent and child. Daily Activity Counts are a measure of frequency and intensity of physical activity, converted from raw acceleration data to unitless count data.
Wearable sensor physical activity data: Average Resting Heart Rate | From enrollment to end of 8-week treatment period
  Wearable sensor outcomes measured in parent and child., Average resting heart rate, measure in beats per minute, provides a measure of cardiorespiratory fitness.
Wearable sensor physical activity data | From enrollment to end of 8-week treatment period
  Wearable sensor outcomes measured in parent and child. Daily sedentary time, measured in minutes, quantifies the amount of time per day spent sitting, lying or otherwise stationary.
Sleep wearable sensor data: total sleep time | From enrollment until end of treatment period ( 8 weeks)
  Sleep data measured in child only. Total sleep time is the amount of time, in minutes, that the child is sleeping.
Sleep wearable sensor data: Sleep Latency | From enrollment until end of treatment period ( 8 weeks)
  Sleep data measured in child only. Sleep latency is a measure of the time gap between when the child lays down at bedtime until they fall asleep, as measured by the wearable sensor. Sleep latency is measured in minutes.
Sleep wearable sensor data: Sleep efficiency | From enrollment until end of treatment period ( 8 weeks)
  Sleep data measured in child only. Sleep efficiency is the proportion of time in bed that the child is asleep and is reported as a percentage.

SECONDARY OUTCOMES:
CP-CHILD | before and after 8-week intervention
  A parent report measured designs to collect data across 6 domains including Activities of daily living, positioning transferring and mobility, comfort and emotions, communication social interaction, health, and overall quality of life. There are a total of 37 questions and. The questionnaire takes between 20 and 30 minutes to complete using a paper or electronic form.
Young Child-Participation in Environment Measure (YC-PEM) | Before and after 8-week treatment
  A parent report measure that provides detailed information about the child's participation home school and in the community. These activities are measured according to frequency, level of involvement, desire for change in child's level of participation, and environmental supports. The YC-PEM includes 28 items and is valid in children 0-5 years old.
The Early Activity Scale for Endurance (EASE) | Before and after 8 week treatment
  Measures endurance during physical activity in children with cerebral palsy. Eleven questions are rated on a 5 point Likert scale with a higher total score indicating higher endurance.
Perceived Stress Scale-14 (PSS-14) | Before and after 8-week treatment period
  Parents rate their stress levels over the past month. Fourteen items are rated on a 5-point Likert scale; higher scores indicate greater perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Heathcock, PhD, Principal Investigator — Ohio State University
Locations (1):
- Pediatric Assessment and Rehabilitation Lab, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided